CLINICAL TRIAL: NCT03241745
Title: Phase II Trial of Single-Agent Nivolumab in Patients With Microsatellite Unstable/Mismatch Repair Deficient/Hypermutated Uterine Cancer
Brief Title: A Study of Nivolumab in Selected Uterine Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-180
Record Dates: First submitted 2017-08-03; First posted 2017-08-07 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Uterine Cancer; Endometrial Carcinoma; Carcinosarcoma; Leiomyosarcoma; Undifferentiated Sarcoma; High Grade Endometrial Stromal Sarcoma; Clear Cell Carcinoma
Keywords: Nivolumab; 17-180
MeSH Terms: conditions — Uterine Neoplasms; Endometrial Neoplasms; Carcinosarcoma; Leiomyosarcoma; Adenocarcinoma, Clear Cell | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: This is an MSKCC investigator-initiated, single-center, non-randomized, open-label, phase 2 study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab treatment: Nivolumab 480 mg IV once every 4 weeks. Treatment will continue until time of disease progression or until development of unacceptable toxicity, whichever comes first.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 480 mg IV once every 4 weeks

SUMMARY:
The purpose of this study is to test the safety of nivolumab and find out what affects, if any, nivolumab has on people and their risk of gynecologic cancer. The investigators also want to find out what effects, good or bad, nivolumab has on the patient and their cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of metastatic or recurrent uterine cancer (endometrial carcinoma, carcinosarcoma, clear cell carcinoma, leiomyosarcoma, undifferentiated sarcoma, high grade endometrial stromal sarcoma) by Memorial Sloan Kettering Cancer Center. Carcinosarcomas, endometrioid and clear cell carcinomas that appears to have arisen in the ovary/fallopian tube or peritoneum are also eligible. Recurrence should not be amenable to curative approaches such as surgical resection or chemoradiotherapy.
* Tumor is confirmed to be one of the following: 1. MSI-high, or 2. MMR-deficient, or 3. Hypermutated defined as ≥20 somatic mutations in the tumor by MSK-IMPACT
* One or more prior lines of cytotoxic treatment for advanced disease (prior hormonal therapy is not considered to count as prior lines of therapy)
* Measurable disease by RECIST 1.1 criteria
* No known CNS metastases
* ECOG Performance status 0-1
* ECOG Performance status 0-1
* WBC ≥ 2000/uL, ANC ≥ 1500/uL, PLT ≥ 100,000/uL, HGB ≥ 8 g/dL
* Serum creatinine ≤ 1.5 x ULN or creatinine clearance of ≥ 40mL/min by Cockroft-Gault formula
* AST (SGOT) and ALT (SGPT) ≤ 3 x ULN
* Total bilirubin ≤ 1.5 x ULN, except subjects with Gilbert's syndrome who can have total bilirubin ≤ 3.0 mg/dL
* Able to sign voluntary written informed consent
* Female, 18 years of age or older
* Available archival tumor tissue or patient is willing to undergo new biopsy
* Premenopausal women of child bearing potential must have a normal urine or serum beta-HCG prior to enrollment, and must agree to use effective contraception during treatment with nivolumab and for at least 5 months following the last dose of nivolumab.

Exclusion Criteria:

* Disease eligible for potentially curative treatment with standard chemotherapy, surgical resection, or chemoradiotherapy.
* Known or suspected autoimmune disease, except for subjects with vitiligo, diabetes mellitus, resolved childhood asthma/atopy, residual hypothyroidism due to an autoimmune immune condition only requiring thyroid hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Serious uncontrolled medical disorder or active infection which would impair the ability of the subject to receive protocol therapy or whose control would be jeopardized by protocol therapy
* History of bowel obstruction, refractory ascites, or bowel perforation due to advanced disease within the past 3 months from start of study treatment.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-CTLA-4 antibody or any other antibody or drug specifically targeting T cell co-stimulation or immune checkpoint pathways
* Patients who have a condition that requires systemic treatment with either corticosteroids within 7 days of enrollment (systemic corticosteroid therapy is defined as >10 mg daily prednisone or its equivalent); or who require other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Prior history of malignancy or a concurrent malignancy, with the exception of cutaneous basal cell carcinoma or squamous cell carcinoma, superficial bladder cancer, or in situ carcinoma of the uterine cervix, prostate, or breast, unless a complete remission was achieved at least 3 years prior to study entry and no additional therapy is required or anticipated to be required during the study period
* Breastfeeding women, pregnant women
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness

  * Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection (if patient has documented Hepatitis B and C from within 6 months of enrollment, these tests do not need to be repeated.)
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Known allergy or Adverse Drug Reaction to nivolumab, or a history of allergy to study drug components.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 35 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Friedman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Friedman CF, Manning-Geist BL, Zhou Q, Soumerai T, Holland A, Da Cruz Paula A, Green H, Ozsoy MA, Iasonos A, Hollmann T, Leitao MM Jr, Mueller JJ, Makker V, Tew WP, O'Cearbhaill RE, Liu YL, Rubinstein MM, Troso-Sandoval T, Lichtman SM, Schram A, Kyi C, Grisham RN, Causa Andrieu P, Wherry EJ, Aghajanian C, Weigelt B, Hensley ML, Zamarin D. Nivolumab for mismatch-repair-deficient or hypermutated gynecologic cancers: a phase 2 trial with biomarker analyses. Nat Med. 2024 May;30(5):1330-1338. doi: 10.1038/s41591-024-02942-7. Epub 2024 Apr 23. PMID 38653864
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab
Started | 35
Completed | 6
Not Completed | 29
Not completed — Adverse Event | 7
Not completed — Death | 1
Not completed — Withdrawal by Subject | 5
Not completed — Treatment delay >28 days | 2
Not completed — Lack of Efficacy | 14

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 64 [36 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 27
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)
Time Frame: at 24 weeks
Measure: Number (97.5% Confidence Interval); unit: percentage of patients
Arm/Group | Nivolumab
Number analyzed (Participants) | 35
percentage of patients | 64.7 [46.5 to 100]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Nivolumab
All-Cause Mortality (participants affected / at risk) | 14/35
Serious Adverse Events (participants affected / at risk) | 12/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=35)
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Acute optic neuritis (Eye disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Atrioventricular Block Complete (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Blood bilirubin increased (Investigations) | 1
Cognitive disturbance (Nervous system disorders) | 1
Creatinine increased (Investigations) | 1
Device related infection (Infections and infestations) | 1
Dizziness (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fever (General disorders) | 1
Hemolysis (Blood and lymphatic system disorders) | 1
Myocarditis (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain (General disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Thromboembolic Event (Vascular disorders) | 3
Urinary tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=35)
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 9
Acute kidney injury (Renal and urinary disorders) | 1
Acute optic neuritis (Eye disorders) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 3
Allergic reaction (Immune system disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3
Anemia (Blood and lymphatic system disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Ascites (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 3
Atrioventricular block complete (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bleeding from gums (Infections and infestations) | 1
Bloating (Gastrointestinal disorders) | 1
Blood bilirubin increased (Investigations) | 1
Blurred vision (Eye disorders) | 3
Breast pain (Reproductive system and breast disorders) | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
C. Difficile (Infections and infestations) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 2
Cognitive disturbance (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 9
Corneal ulcer (Eye disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
COVID 19 (Infections and infestations) | 2
Creatinine increased (Investigations) | 2
Cyst in Left Shoulder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depression (Psychiatric disorders) | 4
Dermatitis radiation (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Diarrhea (Gastrointestinal disorders) | 13
Dizziness (Nervous system disorders) | 8
Dry eye (Eye disorders) | 1
Dry mouth (Gastrointestinal disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 4
Dysgeusia (Nervous system disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
Edema limbs (General disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Extraocular muscle paresis (Eye disorders) | 1
Fall (Injury, poisoning and procedural complications) | 5
Fatigue (General disorders) | 15
Fever (General disorders) | 9
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Flu like symptoms (General disorders) | 1
Renal and urinary disorders - Other, specify (frequency) (Renal and urinary disorders) | 1
Gait disturbance (General disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal pain (Gastrointestinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 7
Hearing impaired (Ear and labyrinth disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hemolysis (Blood and lymphatic system disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Herpes Zoster (no open vesicles) (Infections and infestations) | 1
Hot flashes (Vascular disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypertension (Vascular disorders) | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Investigations) | 5
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 2
Hypothyroidism (Endocrine disorders) | 3
Insomnia (Psychiatric disorders) | 3
Keratitis (Eye disorders) | 1
Leg cramps (Musculoskeletal and connective tissue disorders) | 1
Lip infection (Infections and infestations) | 1
Lipase increased (Investigations) | 3
Localized edema (General disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Lymphedema (Vascular disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Malaise (General disorders) | 2
Memory impairment (Nervous system disorders) | 3
Mucosal infection (Infections and infestations) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Myocarditis (Cardiac disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Nausea (Gastrointestinal disorders) | 17
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Overactive Bladder (Infections and infestations) | 1
Pain (General disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 4
Pharyngitis (Infections and infestations) | 1
Photophobia (Eye disorders) | 1
Pneumonitis (Reproductive system and breast disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 11
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Rectal hemorrhage (Gastrointestinal disorders) | 2
Renal calculi (Renal and urinary disorders) | 1
Retinal vascular disorder (Eye disorders) | 1
Serum amylase increased (Investigations) | 1
Shingles (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Skin infection (Infections and infestations) | 3
Small intestinal obstruction (Gastrointestinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Thromboembolic event (Vascular disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 2
Tremor (Nervous system disorders) | 1
Type 1 Diabetes (Endocrine disorders) | 1
Upper respiratory infection (Infections and infestations) | 6
Urinary frequency (Renal and urinary disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 6
Urinary tract obstruction (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 3
Vaginal discharge (Reproductive system and breast disorders) | 2
Vaginal dryness (Reproductive system and breast disorders) | 4
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Vaginal infection (Infections and infestations) | 2
Vaginal inflammation (Reproductive system and breast disorders) | 1
Vaginal pain (Reproductive system and breast disorders) | 1
Vomiting (Gastrointestinal disorders) | 11
Weight gain (Investigations) | 2
Weight loss (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT03241745/Prot_SAP_000.pdf